CLINICAL TRIAL: NCT00223860
Title: Provocative Testing Using LHRH and hCG of the Pituitary-Gonadal Axis in Persons With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Bauman, William - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B2648
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-03

CONDITIONS: Hypogonadism; Spinal Cord Injury
Keywords: Hypogonadal; Hypothalamus; Pituitary; Spinal Cord Injury; Testes; Testosterone
MeSH Terms: conditions — Hypogonadism; Spinal Cord Injuries; Pituitary Diseases | interventions — Chorionic Gonadotropin; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Human chorionic gonadotropin (hCG); Drug: Luteinizing hormone releasing hormone (LHRH)

INTERVENTIONS:
Drug: Human chorionic gonadotropin (hCG)
Drug: Luteinizing hormone releasing hormone (LHRH)

SUMMARY:
There is evidence that has shown that serum testosterone levels are low in persons with chronic spinal cord injury (SCI). The question arises as to whether the defect in testosterone production is from the hypothalamic pituitary system (part of the brain that plays a role in testosterone release) or from the male testes. Studies to date are inconclusive. This study, will examine if persons with SCI has a normal hormonal regulation of the male hormone testosterone in comparison to persons who are able-bodied. This will help understand the physical and metabolic changes that occur in persons with SCI.

DETAILED DESCRIPTION:
Absolute or relative testosterone deficiency is associated with loss of lean body tissue and gain of fat, with associated adverse carbohydrate, lipid, and energy expenditure changes that increase the risk of cardiovascular disease. Impotence and infertility are common in patients with SCI. Of the many possible explanations of poor semen quality, one possible etiology is dysfunction of the hypothalamic-pituitary-testicular axis. Early reports have been inconclusive with regard to testicular function. These apparent discrepancies could, at least in part, be attributed to varying factors in population selection, including health and nutrition parameters, medication effects, and level and duration of injury, or to differences in methodology. Recently, two large population studies found a sizeable proportion of persons with SCI having testosterone deficiency. Huang et al. (1993) found significantly elevated luteinizing hormone (LH) responses to LH releasing hormone (LHRH) in subjects with SCI compared to controls. Of those studied with LHRH stimulation, 16/30 subjects with SCI had exaggerated LH responses and 6/30 had elevated follicular stimulation hormone (FSH) responses. Bulat et al., (1995) have shown that persons with tetraplegia tend to have increased gonadotropin release to standard provocative stimulation compared with able-bodied controls or those with paraplegia. In a preliminary report, testicular stimulation with standard doses of hCG for 2 days was similar in 10 subjects with SCI and 8 able-bodied controls.

ELIGIBILITY:
Inclusion Criteria:

1. SCI with serum total testosterone 3.0 ng/ml (SCI eugonadal, n=25),
2. SCI with serum total testosterone <3.0 ng/ml (SCI hypogonadal, n=25),
3. able-bodied controls with serum total testosterone 3.0 ng/ml (control eugonadal, n=25), and
4. able-bodied controls with serum total testosterone <3.0 ng/ml (control hypogonadal, n=25). All SCI and control subjects will be screened for serum gonadotropin levels within the normal range as an inclusion criterion.

Exclusion Criteria:

1. acute illness,
2. active thyroid disease,
3. pyschotropic medications,
4. anti-hypertensive medications (centrally acting, i.e., guanethidine, reserpine, methyldopa, b-adrenergic blockers, clonidine, etc.),
5. H2-blockers,
6. digoxin,
7. alcoholism,
8. anti-convulsant medications (dilantin or barbiturates)
9. diuretics (thiazides or spironolactone),
10. chemotherapeutic agents,
11. antibiotics,
12. opiates,
13. hormones (other than replacement doses),
14. history of pituitary or testicular surgery. Abstinence from alcoholic beverages will be required for 48 hours prior to study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2001-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Bauman, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States

REFERENCES:
- [Result] Tsitouras PD, Zhong YG, Spungen AM, Bauman WA. Serum testosterone and growth hormone/insulin-like growth factor-I in adults with spinal cord injury. Horm Metab Res. 1995 Jun;27(6):287-92. doi: 10.1055/s-2007-979961. PMID 7557841
- [Result] Huang TS, Wang YH, Chiang HS, Lien YN. Pituitary-testicular and pituitary-thyroid axes in spinal cord-injured males. Metabolism. 1993 Apr;42(4):516-21. doi: 10.1016/0026-0495(93)90112-2. PMID 8487676
- See also: Click here for more information about this study: Provocative Testing Using LHRH and hCG of the Pituitary-Gonadal Axis in Persons With Spinal Cord Injury — http://www.unitedspinal.org